CLINICAL TRIAL: NCT04185857
Title: Effects of Mineralocorticoid and AT-1 Receptor Antagonism on the Aldosterone-Renin Ratio (ARR) In Primary Aldosteronism Patients (EMIRA Study): Rationale and Design
Brief Title: MRA and ARB Treatment in Screening of Primary Aldosteronism
Acronym: EMIRA
Status: Completed | Type: Observational
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Gian Paolo Rossi, MD, FAHA, FACC, Professor, University Hospital Padova
Other Study IDs: EMIRA-64140
Record Dates: First submitted 2019-11-25; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Primary Aldosteronism Due to Aldosterone Producing Adenoma
Keywords: renin; aldosterone; aldosterone to renin ratio
MeSH Terms: interventions — Canrenone; olmesartan

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients with primary aldosteronism (PA): After two biochemical and clinical evaluations under baseline conditions PA patients will be treated with canrenone 50-100 mg orally once a day.
  After one month of such therapy they will undergo the a clinical and biochemical evaluation (FW1). After, they will continue with a combination therapy with canrenone, plus olmesartan starting with 10 mg a day for oral administration, a dose that can be doubled, if necessary, to achieve normotension.
  At the end of the second month of the double therapy, patients will undergo a biochemical re-evaluation at the Center of Hypertension (FW2).
  Interventions: Drug: canrenone 50-100 mg orally once a day; Drug: olmesartan 10-20 mg orally once a day

INTERVENTIONS:
Drug: canrenone 50-100 mg orally once a day — After two biochemical and clinical evaluations under baseline conditions and after pharmacological washout from diuretics, betablockers, ARBs or ACEI (about 4 weeks) and MRAs (abut 6 weeks), PA patients will be treated with canrenone 50-100 mg orally once a day. After 1 or 2 weeks the dose will be doubled if necessary to control BP and serum potassium.
Drug: olmesartan 10-20 mg orally once a day — After one month of treatment with canrenone the patients will undergo a clinical and biochemical evaluation (FW1) in a manner identical to the two basal evaluations. After, they will continue with a combination therapy with canrenone, at the dose reached, plus olmesartan starting with 10 mg a day for oral administration, a dose that could be doubled, if necessary, to achieve normotension.
  At the end of the second month of the double therapy, patients will undergo a biochemical re-evaluation at the Center of Hypertension (FW2) with methods identical to those performed in the two baseline evaluations and after one month of canrenone.

SUMMARY:
Current guidelines recommend withdrawal of treatments that affect the aldosterone/renin ratio (ARR) when screening for primary aldosteronism (PA). However, abandonment of mineralocorti-coid-receptor antagonist (MRA) and/or blockers of the renin-angiotensin system can deteriorate control of blood pressure (BP) and hypokalemia. Thus, in consecutive patients with an unambiguous diagnosis of PA in wash-out from confounding treatments and subtyped by AVS, the investigators have compared within-patient the plasma aldosterone and active renin concentration, and the ARR values, measured at baseline, and after a one-month treatment with MRA alone and combined with an AT-1 receptor blocker (ARB). Patients on a regular salt intake have been treated with canrenone (50-100 mg orally) for 1 month, after which olmesartan (10 or 20 mg orally) has been added for another month with up-titration of both treatments over the first 2 weeks to control BP and hypokalemia, however maintaining background therapy. The biochemical variables and the ARR have been assessed in an identical manner at baseline values and after each month of treatment. The investigators calculated that with a sample size of 40 patients the study will have a 95% power to show a clinically significant 20% change in the ARR at an 5% alfa-value using a two-sided paired t-test. Hence, this study will allow to determine if an MRA alone, or added to an ARB at doses that control BP and hypokalemia, affect or not the ARR, thus allow to establish if these agents can be administered or must be forbidden during the screening of PA.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is a common form of hypertension caused by aldosterone secretion inappropriate for blood pressure (BP) and volume status. It involves over 11% of the patients referred to specialized hypertension centres, about one fifth of those with drug-resistant hypertension and even a large proportion of the hypertensive patients seen in general practice. The only main subtype of PA that can be unambiguously diagnosed based on post-adrenalectomy using a "five corners" approach is aldosterone-producing adenoma (APA).

In patients undergoing screening for PA the current guidelines recommend pharmacological wash-out or, more correctly, switch to antihypertensive therapy not influencing the values of plasma aldosterone concentration (PAC) and direct renin concentration (DRC) and therefore of the aldosterone/renin ratio (ARR). This therapy generally entails a long-acting calcium channel blocker, alone or in combination with an alpha-blocker. However, a significant proportion of hypertensive patients, about one third, require more complex therapies to maintain acceptable BP levels. In addition, a proportion, estimated at around 10% of patients with PA, have hypertension resistant to common antihypertensives, as shown in the PATWAY-2 study. Noteworthy, these patients usually exibit a BP lowering response to mineralocorticoid-receptor antagonists (MRAs).

MRAs act as diuretics and therefore stimulate the renin-angiotensin-aldosterone system (RAAS), which might confound the results of the diagnostic tests, increasing renin and therefore reducing the ARR. This is considered to increase the rate of false negative tests. Moreover, some data suggest that MRA could inhibit the synthesis of aldosterone. However, this remains contentious as there are no prospective studies in this regard. Therefore, the use of MRAs, which can effectively control BP and hypokalemia during the PA screening is generally discouraged, despite the lack of solid prospective studies in this regard.

The stimulation of SRAA, if it actually occurs in a patient with PA, could be controlled, or prevented, by the use of an angiotensin AT-1 receptor blocker.

Therefore, the investigators set out a prospective observational study aimed at investigating, with a within-patient comparison, the values of PAC, DRC, ARR, serum potassium, in addition to blood pressure, in patients unambigously diagnosed with PA, who underwent screening and subtyping in washout from confounding treatments according to the current guidelines, with the values produced by treatment with MRA (canrenone) given alone or in combination with an angiotensin AT-1 receptor blocker (olmesartan).

Methods:

The investigators will prospectively recruit consecutive PA patients which have been previously studied in washout from confounding treatments (first basal evaluation) and will be subtyped by adrenal vein sampling (AVS) in the Clinica dell'Ipertensione Arteriosa, University of Padova, Italy (second basal evaluation). Inclusion criteria: patients between the ages of 18 and 75, diagnosed with APA according with the guidelines, which will give written informed consent. The exclusion criteria comprise the refusal to participate in the study of the history of intolerance or allergy to canrenone or ARBs.

Patients will be treated with canrenone 50-100 mg orally for 1 month followed by canrenone plus olmesartan 10 or 20 mg for another month. At the end of each month they will undergo a clinical and biochemical reevaluation to investigate the effects of both treatments and compared with the ARR values observed during washout (i.e. during the first and second basal evaluations).

Study design:

After two biochemical and clinical evaluations under baseline conditions and after pharmacological washout from diuretics, betablockers, ARBs or ACEI (about 4 weeks) and MRAs (abut 6 weeks), PA patients will be treated with canrenone 50-100 mg orally once a day. After one and tho weeks the dose will be doubled if necessary to control BP and serum potassium. After one month of such therapy they will undergo the a clinical and biochemical evaluation (FW1) in a manner identical to the two basal evaluations.

After, they will continue with a combination therapy with canrenone, at the dose reached, plus olmesartan starting with 10 mg a day for oral administration, a dose that can be doubled, if necessary, to achieve normotension.

At the end of the second month of the double therapy, patients will undergo a biochemical re-evaluation at the Center of Hypertension (FW2) with methods identical to those performed in the two baseline evaluations and after one month of canrenone.

This protocol is commonly used in the Center of Reference - UOSD Hypertension for the optimal preparation of patients with PA for the eventual intervention of laparoscopic adrenalectomy.

Primary endpoint:

This is a prospective, within-patient, observational study aiming at comparing, in patients with PA, the values of PAC, DRC and ARR assessed in wash-out (or in treatment with CCBs and or alfa-blockers) with the values observed after 1 month treatment with canrenone 50 or 100 mg o.d. and after another month treatment with canrenone 50 or 100 mg o.d. plus olmesartan 10 mg or 20 mg o.d.

Sample size calculation and statistical analysis A statistical power to detect any intra-patient difference of ormonal concentrations will be reached considering 40 patients.

The analysis of the data will be performed initially globally (i.e. on the entire cohort) and subsequently conducted separately: in patients with APA where the diagnosis will be confirmed at the adrenalectomy and biochemical follow-up one month after surgery, and in patients with PA not lateralized where the one month follow up will be performed.

Expected Results. The investigators expect to conclusively determine if and how MRA alone or combined with an ARB at doses that control BP and hypokalemia, affect plasma concentration of PAC and DRC and therefore the ARR.

If the results of this study will not show a confounding effect of one or the other treatment, this study could open the way to perform the screening tests for PA without the need to suspend these treatments and therefore with the possibility of minimizing the risks due to the reduction of therapy antihypertensive in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 75 years;
* diagnosis of Aldosterone Producing Adenoma (APA);
* written informed consent.

Exclusion Criteria:

* refusal to participate to the study;
* history of intolerance or allergy to canrenone or ARB.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive PA patients subtyped with adrenal vein sampling (AVS) at the University of Padova, Italy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Aldosterone to renin ratio (ARR) | one month
  ARR measured as ng/mIU after treatment with canrenone, or olmesartan on top of canrenone

SECONDARY OUTCOMES:
Serum potassium levels | one month
  Serum potassium measured as mmol/L after treatment with canrenone, or olmesartan on top of canrenone
Blood pressure | one month
  Blood pressure measured as mmol/L after treatment with canrenone, or olmesartan on top of canrenone

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Rossi, Study Director — University of Padova
Locations (1):
- Department of Medicine - DIMED, University of Padova, Italy, Padua, Italy

REFERENCES:
- [Result] Rossitto G, Cesari M, Ceolotto G, Maiolino G, Seccia TM, Rossi GP. Effects of mineralocorticoid and AT-1 receptor antagonism on the aldosterone-renin ratio (ARR) in primary aldosteronism patients (EMIRA Study): rationale and design. J Hum Hypertens. 2019 Feb;33(2):167-171. doi: 10.1038/s41371-018-0139-x. Epub 2018 Dec 5. PMID 30518805
- [Result] Rossi GP, Bernini G, Caliumi C, Desideri G, Fabris B, Ferri C, Ganzaroli C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Mattarello MJ, Moretti A, Palumbo G, Parenti G, Porteri E, Semplicini A, Rizzoni D, Rossi E, Boscaro M, Pessina AC, Mantero F; PAPY Study Investigators. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. J Am Coll Cardiol. 2006 Dec 5;48(11):2293-300. doi: 10.1016/j.jacc.2006.07.059. Epub 2006 Nov 13. PMID 17161262
- [Result] Douma S, Petidis K, Doumas M, Papaefthimiou P, Triantafyllou A, Kartali N, Papadopoulos N, Vogiatzis K, Zamboulis C. Prevalence of primary hyperaldosteronism in resistant hypertension: a retrospective observational study. Lancet. 2008 Jun 7;371(9628):1921-6. doi: 10.1016/S0140-6736(08)60834-X. PMID 18539224
- [Result] Seccia TM, Caroccia B, Gomez-Sanchez EP, Gomez-Sanchez CE, Rossi GP. The Biology of Normal Zona Glomerulosa and Aldosterone-Producing Adenoma: Pathological Implications. Endocr Rev. 2018 Dec 1;39(6):1029-1056. doi: 10.1210/er.2018-00060. PMID 30007283
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393